CLINICAL TRIAL: NCT01287312
Title: Trichloroacetic Acid for Endoscopic Tracho-esophageal Fistula Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Shlomo Cohen, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: shlomoco-HMO-CTIL
Record Dates: First submitted 2011-01-27; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Tracheo Esophageal Fistula
Keywords: We will treat children age 1 month to 20 years with recurrent TEF after surgical failure
MeSH Terms: conditions — Tracheoesophageal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic repair of recurrent TEF by trichloroacetic acid aplications

SUMMARY:
Today Endoscopic repair of recurrent Tracheesophageal fistula (TEF) is a safe procedure. Using Trichlosiacetic acid 50% (TCA) for endoscopic aplication of the fistula was reported with a good results ( 4 cases). There were no serious advers effects.

The investigators want to use also TCA 50% for endoscopic repair in children with recurrent TEF.

DETAILED DESCRIPTION:
Today Endoscopic repair of recurrent Tracheesophageal fistula (TEF) is a safe procedure. Using Trichlosiacetic acid 50% (TCA) for endoscopic aplication of the fistula was reported with a good results ( 4 cases). There were no serious advers effects.

We want to use also TCA 50% for endoscopic repair in children with recurrent TEF.

ELIGIBILITY:
Inclusion Criteria:

* children age 1 month- 20 years old with recurrent TEF.
* Failure of surgical repair.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Closure of the fistula
  Closure of the fistula

SECONDARY OUTCOMES:
clinical and pulmonary improvment

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel